CLINICAL TRIAL: NCT02072642
Title: Light Therapy in Parkinson's Disease : Effect on Motor Symptoms, Sleep, Circadian Rhythms, and Mood
Brief Title: Light Therapy in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5063
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active light therapy (10,000 lux) (Active Comparator): Light therapy: DayVia lamp 10000 lux
  Interventions: Device: active light therapy : Light therapy: DayVia lamp 10000 lux
- Placebo light therapy (70 lux) (Placebo Comparator): Placebo light therapy
  Interventions: Device: Placebo light therapy

INTERVENTIONS:
Device: active light therapy : Light therapy: DayVia lamp 10000 lux — 4 weeks of active light therapy with DayVia lamp 10000 lux
  Arms: Active light therapy (10,000 lux)
Device: Placebo light therapy — 4 weeks with Placebo light therapy
  Arms: Placebo light therapy (70 lux)

SUMMARY:
Parkinson's disease, a degenerative disorder of the dopaminergic system, combines motor symptoms but also non-motor, such as depression, sleep disorders and circadian rhythms and impaired cognitive functions. Difficulties in balancing the dopaminergic treatment of these patients emphasizes the need to find effective adjuvant therapies. Light therapy (LT) represents one such innovative therapeutic approach. Although light has an obvious to visual pathways within the brain, today it is known to additionally exert non-visual effects throughout the body. Recently our team has shown that non-visual, non-circadian light plays a major role in the regulation of sleep, as well as cognitive brain function in general. The retina, the primary conduit for the transmission of light information is weakened or thinned in Parkinson's patients. The dopamine system is known to enhance the processing of light information and intraocular injection of L-dopa in animal models of Parkinson's disease, can reverse associated motor symptoms. This allows for the possibility that LT would strengthen the dopaminergic tone in the central nervous system. However, to this date its effectiveness for alleviating Parkinson's symptoms has only been suggested by two studies, both poorly controlled. Thus, through the convergence of basic and clinical data, a study examining the effect of LT directly in people Parkinson's disease symptoms, whilst controlling for the effects on sleep, circadian system, mood, and cognitive functioning, is of extreme importance. With this information our hope is to determine if these polymorphisms allow for a predictive model of response to LT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkison's Disease, low or moderately severe
* Hoehn&Yahr <4
* 4 to < 15 years of evolution·
* Between 45-75 years old
* Absence of dementia : MMSE > 23·
* No severe depression
* Stable medication levels during the 5 weeks before inclusion

Exclusion Criteria:

* Secondary or severe Parkinson's disease
* Ocular pathologies (i.e. retinopathy)
* Photosensitive medication
* Antidepressant treatment·
* Major depression syndrome
* MMSE < 23
* Circadian rhythm problems
* Sleep apnea syndrome
* Manifested or acute psychiatric comorbidities
* Pregnant women

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Global score :Unified Parkinson's Disease Rating Scale (UPDRS) I II III | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrice BOURGIN, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No